CLINICAL TRIAL: NCT01052701
Title: Pharmacokinetic Interactions of Ribavirin and Abacavir in Hepatitis-C Mono-infected Male Subjects Who Previously Failed Ribavirin-based Treatment
Brief Title: Drug Interaction Study With Ribavirin and Abacavir in Male Subjects With Hepatitis C Who Have Failed Ribavirin Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: GlaxoSmithKline (Industry); University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NA_00023807
Record Dates: First submitted 2010-01-19; First posted 2010-01-20 (Estimated); Results first posted 2017-04-27 (Actual); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Hepatitis C; HIV
MeSH Terms: conditions — Hepatitis C | interventions — Ribavirin; abacavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ribavirin plus Abacavir (Active Comparator): Ribavirin plus Abacavir Administration intervention
  Interventions: Drug: Ribavirin plus Abacavir (ABC)
- Ribavirin alone (Active Comparator): Ribavirin alone administration
  Interventions: Drug: Ribavirin

INTERVENTIONS:
Drug: Ribavirin — Daily Ribavirin alone 400 mg in the morning (AM) and 600 mg in the afternoon (PM) orally with 12 hours between the doses (Body Weight ≤75 kg)
  OR
  Daily RBV alone 600 mg orally every 12 hours (Body Weight >75 kg)
  Other Names: Ribavirin (RBV)
  Arms: Ribavirin alone
Drug: Ribavirin plus Abacavir (ABC) — Daily Ribavirin 400 mg in AM and 600 mg in PM orally with 12 hours between the doses (Body Weight ≤75 kg)
  OR
  Daily RBV 600 mg orally every 12 hours (Body Weight >75 kg)
  Plus
  Daily Abacavir 300 mg orally every 12 hours
  Other Names: RBV + ABC
  Arms: Ribavirin plus Abacavir

SUMMARY:
This research is being done to find out whether abacavir (Ziagen®) lowers the levels of ribavirin (Ribapak®) in the body of persons taking these two drugs.

DETAILED DESCRIPTION:
Abacavir is an anti-HIV drug that belongs to the class of nucleoside reverse transcriptase inhibitors. Ribavirin is a drug used to treat hepatitis C infection. Both abacavir and ribavirin are approved by the Food and Drug administration (FDA). The doses of abacavir and ribavirin used in this study are also FDA approved.Some individuals who have HIV infection also have hepatitis C. It is possible that they may need to take both abacavir to treat HIV and ribavirin to treat hepatitis C. Recent studies suggest that abacavir decreases the level of ribavirin in the body, in the blood and in cells named peripheral blood mononuclear cells (PBMC's). Thus, taking ribavirin and abacavir together could lead to treatment failure for hepatitis C. Therefore, it is important to understand whether ribavirin levels are affected when the two medications are taken together.

ELIGIBILITY:
Inclusion Criteria:

* Hepatitis C Virus (HCV) -monoinfected subjects who either successfully completed (defined as cured) or previously failed RBV-based therapy for hepatitis C infection, and are currently not receiving therapy for hepatitis C; at least 18-64 years of age. HCV cure is defined as a sustained undetectable viral response at 24 weeks post treatment.
* Females who are not of reproductive potential (defined as women who have been postmenopausal for at least 24 consecutive months or who have undergone hysterectomy, bilateral oophorectomy, or bilateral tubal ligation.
* Negative serum β- human chorionic gonadotropin (HCG)
* Negative HIV-1 serology documented by any licensed Enzyme-linked immunoassay (ELISA) test kit within 30 days prior to study entry.
* Positive HCV antibody documented within 30 days prior to study entry.
* Negative Human Leukocyte Antigen (HLA)-B*5701 test documented within 30 days prior to study entry.
* Ability and willingness of subject to provide a signed informed consent and comply with study requirements.
* All subjects must not participate in a conception process (e.g., active attempt to impregnate, sperm donation, in vitro fertilization). If participating in sexual activity that could lead to pregnancy, male subjects must take every precaution to avoid risk of pregnancy for their female partners by using reliable contraception (condom) while receiving study therapy and for 6 months following permanent discontinuation of study therapy. Subjects will also be instructed to counsel their female partners regarding fetal risk and need for appropriate contraception (e.g., hormonal, barrier) so as a secondary effort to prevent pregnancy even though the female partners will not be study participants.
* Estimated creatinine clearance ≥50 mL/minute, within 30 days prior to study entry
* Laboratory values obtained within 30 days prior to study entry:
* Hgb within the normal limits as defined by the reporting laboratory
* Aspartate aminotransferase (AST), Alanine aminotransferase (ALT), and alkaline phosphatase >5 x upper limit of normal (ULN) as defined by the reporting laboratory.
* Direct bilirubin ≤1.5 x ULN as defined by the reporting laboratory.
* Follicle Stimulate Hormone (FSH) measurement elevated into the menopausal range for females who report being postmenopausal for at least 24 consecutive months is required at screening for all female subjects.
* Subject has not consumed alcohol in the 48 hours prior to the administration of study drugs.
* Framingham cardiovascular disease risk score <10%.

Exclusion Criteria:

* As determined by the investigator, a significant active or previous history of cardiovascular, renal, hematologic, neurologic, gastrointestinal, psychiatric, endocrine, or immunologic disease (s). This inclusive of chronic illnesses such as hypertension, coronary artery disease, arthritis, diabetes, any chronic gastrointestinal condition that may affect drug absorption. History of chronic or acute medical condition that in the opinion of the investigator would jeopardize safety of subjects participating in this study. Any other medical or psychological condition that might, in the opinion of the site investigator, interfere with participation in the study or put subjects at undue risk.
* History of anemia, hemoglobinopathy or any other cause of or tendency to hemolysis.
* History of RBV-induced anemia that required dose reduction or discontinuation of RBV therapy while receiving treatment for hepatitis C infection in the past. Patients who required treatment with erythropoietin or blood transfusion for the management of RBV-associated anemia will be excluded from participating in the study.
* Use of prescription or over-the-counter medications, including herbal products, within 30 days prior to study entry that in the opinion of the investigator would preclude study participation.
* Pregnant women or men with a pregnant female partner.
* Breast feeding
* Active drug use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements, and/or currently receiving methadone replacement therapy for the treatment of substance abuse.
* Inability of abstaining from alcohol-containing beverages for the duration of the study.
* Hospitalization or therapy for serious illness within 30 days prior to study entry as judged by the investigator.
* Known or suspected hypersensitivity reaction to study drugs or their formulations.
* Participation in any investigational drug study within 30 days prior to study entry.
* Active or history of gout disease.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2009-12; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Andrade, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Drug Development Unit, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fuchs EJ, Kiser JJ, Hendrix CW, Sulkowski M, Radebaugh C, Bushman L, Ray ML, Andrade A. Plasma and intracellular ribavirin concentrations are not significantly altered by abacavir in hepatitis C virus-infected patients. J Antimicrob Chemother. 2016 Jun;71(6):1597-600. doi: 10.1093/jac/dkw009. Epub 2016 Feb 10. PMID 26869690

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited through general newspaper advertisements, flyers, and referral from providers specializing in hepatitis C
Groups:
- Ribavirin Plus Abacavir: Ribavirin plus Abacavir Administration intervention
  Ribavirin plus Abacavir: Daily Ribavirin 400 mg in the morning (AM) and 600 mg in the afternoon (PM) orally with 12 hours between the doses (Body Weight ≤75 kg)
  or
  Daily RBV 600 mg orally every 12 hours (Body Weight >75 kg)
  plus
  Daily Abacavir 300 mg orally every 12 hours
- Ribavirin Alone: Ribavirin alone administration
  Ribavirin: Daily Ribavirin alone 400 mg in AM and 600 mg in PM orally with 12 hours between the doses (Body Weight ≤75 kg)
  OR
  Daily RBV alone 600 mg orally every 12 hours (Body Weight >75 kg)
Period: Overall Study
Arm/Group | Ribavirin Plus Abacavir | Ribavirin Alone
Started | 14 | 12
Completed | 14 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Ribavirin Plus Abacavir: Ribavirin plus Abacavir Administration intervention
  Ribavirin plus Abacavir: Daily Ribavirin 400 mg in AM and 600 mg in PM orally with 12 hours between the doses (Body Weight ≤75 kg)
  or
  Daily RBV 600 mg orally every 12 hours (Body Weight >75 kg)
  plus
  Daily Abacavir 300 mg orally every 12 hours
- Total: Total of all reporting groups
Arm/Group | Ribavirin Plus Abacavir | Ribavirin Alone | Total
Number analyzed (Participants) | 14 | 12 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 12 | 26
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 54 [50 to 58] | 50 [48 to 54] | 52 [49 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 13 | 12 | 25
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 12 | 26

OUTCOME MEASURES:

1. Primary Outcome: Ribavirin Triphosphate (RBV-TP) Intracellular Concentrations
Description: Ribavirin Triphosphate (RBV-TP) intracellular concentrations.
Time Frame: Day 56
Measure: Mean (Standard Deviation); unit: picomoles per 10^6 cells
Arm/Group | Ribavirin Plus Abacavir | Ribavirin Alone
Number analyzed (Participants) | 14 | 12
picomoles per 10^6 cells | 15.87 (12.82) | 15.93 (12.69)

2. Secondary Outcome: Plasma RBV Trough Concentrations
Description: Plasma RBV trough concentrations.
Time Frame: Day 56
Measure: Mean (Standard Deviation); unit: micrograms per milliliter
Arm/Group | Ribavirin Plus Abacavir | Ribavirin Alone
Number analyzed (Participants) | 14 | 12
micrograms per milliliter | 2.54 (1.05) | 2.60 (0.62)

ADVERSE EVENTS:
Arm/Group | Ribavirin Plus Abacavir | Ribavirin Alone
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/12
Other Adverse Events (participants affected / at risk) | 10/14 | 11/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ribavirin Plus Abacavir (N=14) | Ribavirin Alone (N=12)
hyperbilirubinemia (Hepatobiliary disorders) | 2 (2) | 3 (3)
fatigue (General disorders) | 4 (4) | 0 (0)
hyperglycemia (Endocrine disorders) | 10 (10) | 8 (8)
insomnia (General disorders) | 2 (2) | 1 (1)
nausea (Gastrointestinal disorders) | 1 (1) | 3 (3)
transaminitis (Hepatobiliary disorders) | 5 (5) | 4 (4)
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No